CLINICAL TRIAL: NCT01375010
Title: The Effect of Vitamin D Repletion on Postmenopausal Women With HIV
Brief Title: Vitamin D HIV Study on Postmenopausal Women
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Elizabeth Shane, Professor of Medicine, Endocrinology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAAF2194; 2R01AI065200-06A1 (NIH)
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: HIV
Keywords: HIV; Postmenopausal women; Vitamin D
MeSH Terms: interventions — Cholecalciferol; Geritol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Placebo Comparator): Placebo vitamin D3 capsule daily plus vitamin supplements that contains 1000 IU vitamin D3 and 1000 mg calcium carbonate daily. Total daily vitamin D3 dose = 1000 IU.
  Interventions: Other: Placebo; Drug: Vitamin Supplements
- Group B (Experimental): 2000 IU vitamin D3 daily plus vitamin supplements that contains 1000 IU vitamin D3 and 1000 mg calcium carbonate daily. Total daily vitamin D3 dose = 3000 IU.
  Interventions: Drug: Vitamin D3; Drug: Vitamin Supplements

INTERVENTIONS:
Drug: Vitamin D3 — 2000 mg QD
  Other Names: cholecalciferol-D3
  Arms: Group B
Other: Placebo — An inactive treatment that is intended to provide baseline measurements for the experimental protocol of a clinical trial, in this case, the vitamin D3.
  Other Names: Placebo capsule
  Arms: Group A
Drug: Vitamin Supplements — Specially formulated supplements (Tishcon, Inc.) that contain 500 mg of calcium (carbonate) and 500 IU of vitamin D3 to be taken twice daily with breakfast and dinner (1000 mg of elemental calcium and 1000 IU of vitamin D).
  Other Names: Vitamin supplementation

SUMMARY:
The purpose of this study is to determine the effects of vitamin D on measures of bone health and immune function in HIV infected postmenopausal women. The investigators prior research with this population revealed that low vitamin D levels are very common. Prior research with this population also revealed that Vitamin D is necessary for the body to absorb calcium and is important for the health of the bones. When vitamin D levels are low, there are increased risks of bone loss, muscle weakness, falls and fractures. Low levels of vitamin D have also been associated with impaired immune function. This study will help us learn whether two different doses of vitamin D will improve bone health and immune function.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of vitamin D repletion on rates of bone loss and indices of immune function in HIV+ postmenopausal women. Lower baseline serum Vitamin D levels, as assessed by measuring serum 25-hydroxyvitamin D (25-OHD) were associated with a trend toward more bone loss. In addition, the investigators found that despite providing supplements that contained approximately 600 IU vitamin D, serum 25-OHD did not increase during the first year. Provision of adequate calcium and vitamin D is the cornerstone of effective prevention and therapy of osteoporosis. HIV-infected patients may be at increased risk of having vitamin D deficiency because they take several medications that may interfere with vitamin D action. Therefore, the investigators will recruit 100 HIV infected postmenopausal women for this study who are on a stable antiretroviral therapy (ART) regimen and randomize them to receive 1000 or 3000 IU of vitamin D daily. The subjects will be followed closely for one year to monitor compliance and changes in bone health and immune function.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ African American and Latina postmenopausal women, aged 40-70, who meet the standard definition of menopause:

If 50 years old or older then amenorrhea for > 1year. If age 40 to 49 then amenorrhea for over a year and and Follicle-Stimulating Hormone (FSH) level of equal to or greater than 20 mIU/ml; as some amenorrheic chronically ill women may have hypothalamic dysfunction and low FSH values, if FSH is 10 to 19, and the serum estradiol level is consistent with menopause less than or equal to 30pg/ml, she will be determined to be postmenopausal.

* On stable antiretroviral therapy (ART) for >2 years
* Undetectable HIV RNA (viral load) at least 2 times over the past year (RNA <400)

Exclusion Criteria:

* Metabolic bone disease (Paget's disease, clinical osteomalacia, primary hyperparathyroidism, hypercalcemia)
* Multiple myeloma, solid tumors with metastases;
* Endocrinopathy (hyperthyroidism, untreated hypothyroidism, Cushing's syndrome, prolactin-secreting pituitary adenoma)
* Renal insufficiency (serum creatinine above 1.5 mg/dl)
* Liver disease (AST, ALT, bilirubin, total alkaline phosphatase activity > twice upper normal limit);
* Intestinal disorders (celiac disease, pancreatic insufficiency, Crohn's disease, ulcerative colitis)
* Current use of glucocorticoids, anticonvulsants, anticoagulants, diuretics, methotrexate;
* Current or past use of drug therapies for osteoporosis (raloxifene, bisphosphonates, calcitonin, PTH). Women on estrogen are excluded. Past estrogen use is permitted if discontinued >1 year before enrollment.
* If there is a history of a low trauma fracture, a T score < -3 or a prevalent vertebral fracture on Instant Vertebral Assessment™ (IVA), subjects will be referred for osteoporosis treatment as appropriate.
* Severe vitamin D deficiency (25-OHD level <10 ng/ml) or normal baseline serum vitamin D (25-OHD >32 ng/ml). Subjects with severe vitamin D deficiency may be referred to our sub-study, if all other inclusion/exclusion criteria are met.
* Hypercalcemia or history of calcium-containing kidney stones
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulations
* Current imprisonment or voluntary incarceration in a medical facility for psychiatric illness
* Any condition that, in the opinion of the site investigator, would compromised the subject's ability to participate in the study

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Shane, MD, Principal Investigator — Columbia University; Michael Yin, MD, Study Director — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 43 | 42
Completed | 31 | 38
Not Completed | 12 | 4
Not completed — Lost to Follow-up | 8 | 2
Not completed — Withdrawal by Subject | 4 | 2

BASELINE CHARACTERISTICS:
Population: HIV-infected postmenopausal African American or Hispanic women between ages 40-70 were recruited from 4 sites in New York City. All participants had serum 25-OHD ≥10 ng/mL and < 32 ng/mL and were on stable ART for at least 2 years with 2 or more HIV RNA levels <400 copies/ml within the last year prior to enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (4.9) | 56.5 (5.6) | 56.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 85
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 17 | 20 | 37
  Hispanic | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD)
Description: Percent change from baseline in BMD at lumbar spine (as measured by Dual-emission X-ray absorptiometry (DXA) scan) at 12 months
Time Frame: Baseline, 12 months
Population: A complete case approach was utilized for outcome in participants with BMD data at 12 months (n=69).
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 31 | 38
percentage change | 0.4 (4.4) | -0.8 (4.6)

2. Secondary Outcome: Areal Change in Bone Mineral Density (aBMD)
Description: To evaluate the change in areal BMD (aBMD) at the total hip (TH)
Time Frame: Baseline,12 months
Population: A complete case approach was utilized for outcome in participants with BMD data at 12 months (n=69).
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 31 | 38
percentage of change | -0.5 (3.1) | -0.8 (3.2)

3. Secondary Outcome: Change in Volumetric Bone Mineral Density (vBMD)
Description: To evaluate the change in volumetric BMD (VBMD) at the Tibia
Time Frame: Baseline, 12 months
Population: A complete case approach was utilized for secondary outcomes in participants with vBMD data at 12 months (n=69).
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 31 | 38
percentage of change | -0.3 (2.9) | -0.9 (2.5)

4. Secondary Outcome: Change in Vitamin D Levels
Description: To evaluate the change in vitamin D levels with supplementation
Time Frame: 12 months
Population: A complete case approach was utilized for secondary outcomes in participants with data at 12 months (n=69).
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 31 | 38
percentage of change | 33.7 (41.9) | 64.1 (68.6)

5. Secondary Outcome: Change in Biochemical Markers
Description: To evaluate the effect of vitamin D and calcium supplementation on biochemical markers of bone turnover and markers of inflammation. (PTH)
Time Frame: 12 months
Population: A complete case approach was utilized for secondary outcomes in participants with data at 12 months (n=69).
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group A | Group B
Number analyzed (Participants) | 31 | 38
percentage of change | -7.2 (71.4) | -16.8 (33.0)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event reporting was collected at every visit as part of the protocol.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/43 | 1/42
Other Adverse Events (participants affected / at risk) | 6/43 | 5/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=43) | Group B (N=42)
Rectal bleeding/ hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Evidence of internal and external hemorrhoids
Cardiac Ischemia (Cardiac disorders) | 0 (0) | 1 (1) — Infarction
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=43) | Group B (N=42)
Pain (General disorders) | 2 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Kidney Stones (Renal and urinary disorders) | 2 (2) | 3 (3) — Asymptomatic kidney stones at baseline visit scans

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No